CLINICAL TRIAL: NCT05289466
Title: Oncoplastic Partial Mastectomy With Intraoperative Radiation Therapy (IORT) in Early Stage Breast Cancer Patients With Prior History of Chest Wall Radiation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal research admin issue required this study to be closed, will re-open an amended protocol.
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Principal Investigator, Janie Grumley, Director, Margie Petersen Breast Center; Associate Professor of Surgery, Saint John's Cancer Institute, Saint John's Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCI OBCS WITH IORT
Record Dates: First submitted 2022-03-08; First posted 2022-03-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: IORT-Intra-Operative Radiation Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, Non-randomized, Single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-arm (Other): Intraoperative Radiotherapy (Xoft, 20 Gy single dose)
  Interventions: Radiation: Intraoperative Radiotherapy; Procedure: Oncoplastic partial mastectomy

INTERVENTIONS:
Radiation: Intraoperative Radiotherapy — Intraoperative Radiotherapy (Xoft, 20 Gy single dose)
Procedure: Oncoplastic partial mastectomy — Breast Conserving Therapy

SUMMARY:
Prospective, Non-randomized, Single-arm.The objectives of this study are to evaluate cosmesis and perioperative complications associated with the use of intraoperative radiotherapy (IORT) at the time of partial mastectomy in patients with breast cancer and a prior history of radiation therapy. Secondary objectives include evaluating effectiveness of partial mastectomy with IORT, measured by local, regional and distant recurrence, mastectomy rate, and disease-specific and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 y.o.
* Histologically proven in situ and invasive ductal or lobular breast recurrence
* Prior history of whole breast/chest wall radiation therapy
* Disease span ≤ 3 cm, unifocal
* No nodal disease (N0)
* No evidence of metastatic disease (M0)
* Time from initial BCT should be ≥ 1 year
* Patients have refused the standard of care of mastectomy
* Skin distance of ≥ 0.8 cm between applicator and skin

Exclusion Criteria:

* Multifocal and/or multicenter recurrence

  * N1-3 status: Regional cytological or histologically proven node recurrence
  * M1 status: Metastatic disease
  * cT4 (Skin or muscle involvement) or Paget's disease of the nipple
  * Patients undergoing mastectomy
  * Patients undergoing neoadjuvant systemic therapy
  * Connective tissue disease or scleroderma, contraindicating radiotherapy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological Female
Enrollment: 5 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Cosmetic Outcomes as evaluated using BREAST-Q questionnaire as a measure of patient-reported ratings. | 5 years
  The BREAST-Q is a validated patient-reported outcome measure of breast related satisfaction and quality of life, including psychosocial, sexual well-being, and physical domains. Data for cosmetic outcomes will be summarized at the study's completion. This data will be compared to patients included in the IORT Registry that did not have a history of prior irradiation utilizing appropriate statistical tests and models.
Cosmetic Outcomes as evaluated using the Harvard Breast Cosmesis Grading Scale as a measure of patient-reported ratings. | 5 years
  Data for cosmetic outcomes will be summarized at the study's completion. This data will be compared to patients included in the IORT Registry that did not have a history of prior irradiation utilizing appropriate statistical tests and models.
Cosmetic Outcomes as evaluated by clinician completion of the Harvard Breast Cosmesis Grading Scale | 5 years
  Data for cosmetic outcomes will be summarized at the study's completion. This data will be compared to patients included in the IORT Registry that did not have a history of prior irradiation utilizing appropriate statistical tests and models.
Perioperative complications as documented using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (CTCAE.v5) scoring system. | 5 years
  Data for perioperative complications will be summarized at the study's completion. This data will be compared to patients included in the IORT Registry that did not have a history of prior irradiation utilizing appropriate statistical tests and models.

SECONDARY OUTCOMES:
Effectiveness of partial mastectomy with IORT, measured by local recurrence. | 5 years
  Tumor recurrence data will be considered a dichotomous outcome, not a time-to-event outcome.
Effectiveness of partial mastectomy with IORT, measured by regional recurrence. | 5 years
  Tumor recurrence data will be considered a dichotomous outcome, not a time-to-event outcome.
Effectiveness of partial mastectomy with IORT, measured by distant recurrence. | 5 years
  Tumor recurrence data will be considered a dichotomous outcome, not a time-to-event outcome.
Effectiveness of partial mastectomy with IORT, measured by mastectomy rate. | 5 years
  Mastectomy rate will be measured by counting those who receive IORT and whose final pathology shows node positive or multifocal disease span >3cm post IORT, are advised to have mastectomy and have mastectomy.
Effectiveness of partial mastectomy with IORT, measured by disease-specific survival. | 5 years
  Disease specific survival will be measured based on dates and causes of death.
Effectiveness of partial mastectomy with IORT, measured by overall survival | 5 years
  Overall survival will be measured based on dates and causes of death.

CONTACTS AND LOCATIONS:
Overall Officials: Janie L Weng Grumley, MD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- Providence Saint John's Hospital, Santa Monica, California, United States